CLINICAL TRIAL: NCT01750450
Title: Validation of Peripheral Pressure Volume Loops and Ultrasound-derived "Cardiac Power" by Comparison With Invasive Left Ventricular Pressure Volume Loops
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 16494
Record Dates: First submitted 2012-12-06; First posted 2012-12-17 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Disease
Keywords: Pressure Volume Area; Pressure Flow Area; Myocardial Work
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective left heart cath: Patients undergoing elective left heart catheterization will be consented for this study

SUMMARY:
The investigators will generate pressure-flow loops and pressure-volume loops from aortic and left ventricular pressure waveforms and Doppler (desc. aorta) flow waveforms and compare left ventricular to arterial pressure-flow and pressure-volume loops as well as to cardiac power from the USCOM 1A device. The goal of this study is to test the hypothesis that non-invasive estimates of cardiac pressure-volume work (derived from ultrasound-based measurements) correlate with invasive estimates.

DETAILED DESCRIPTION:
Extensive animal work by Suga et al. in the 1980s clearly demonstrate a relationship between left ventricular pressure volume area (PVA) and myocardial consumption of oxygen (MVO2).

PVA can be measured by combining radial artery pressures with ultrasound-derived estimates of aortic blood flow. Because the aorta and peripheral artery compartments are separated from the left ventricle by the aortic valve, the peripheral arterial pressures cannot perfectly approximate left ventricular pressures. However, because the majority of variation in the pressure volume loops is made up of changes in height and width (changes in the left ventricular end-diastolic curve are, by contrast, relatively small), both of which can be readily detected by changes in the peripheral arterial blood pressure tracing, this loss of information may be clinically insignificant.

USCOM, has developed a portable suprasternal Doppler probe (model 1A) capable of estimating left ventricular stroke volume; a unique feature of this device is its ability to utilize both stroke volume, heart rate, and mean arterial pressure in an attempt to measure cardiac power. This device has not been validated against invasive estimates of cardiac power.

Knowledge of MVO2 would be a useful clinical variable but is not widely available. The ability to non-invasively estimate MVO2 intraoperatively would give anesthesiologists the ability to measure the effect of hemodynamic interventions on myocardial consumption of oxygen and, when combined with stroke volume, estimate myocardial efficiency. Non-invasively estimates of MVO2 may also allow cardiologists a novel means of assessing the myocardium of patients with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 or older)
* Undergoing left heart catheterization

Exclusion Criteria:

* Unable to visualize ascending aorta using ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18 and over undergoing elective left heart catheterization
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Correlation between left ventricular pressure volume area (PVA) and aortic PVA | day of procedure
  The primary hypothesis of this study is that the slope of the regression line between left ventricular pressure volume area (PVA, as determined by simultaneous measurement of aortic outflow and left ventricular pressures) and aortic PVA (as determined by simultaneous measurement of aortic outflow and radial artery pressure) is not zero. The null hypothesis is that the probability that the slope of the regression line is different from a line with a slope of 0 is greater than 5%.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States